CLINICAL TRIAL: NCT07317739
Title: SCRiCaViPS Screening and Rehabilitation of Visual Field Defects in Post-Stroke Patients
Brief Title: Screening and Rehabilitation of Visual Field Defects in Post-Stroke Patients
Acronym: SCRiCaViPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione David Chiossone - Impresa Sociale (Other)
Collaborators: IRCCS AOU San Martino, Genova, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SCRiCaViPS
Record Dates: First submitted 2025-12-04; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hemianopia; Visual Field Defect Following Cerebrovascular Accident
Keywords: Post stroke visual defects; Screening; Visual field; Rehabilitation; Neurorehabilitation; visual-auditory stimulation
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Intervention Model Description: Study type: interventional. Allocation: randomized Intervention model: parallel assignment (1:1) This study involves two treatment groups of post-stroke patients with visual field defects identified during the screening activity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard intervention (Other): This group of patients will continue according to current clinical practice (control group), directed towards possible neuro-motor rehabilitation until full recovery, and will have access to visual rehabilitation following full recovery of physical condition.
  The follow up visual field test will detect the percentage of spontaneous recovery of the visual field defect during the observation period
  Interventions: Diagnostic Test: Early visual field test
- Early intervention rehabilitation (Experimental): The experimental group will be enrolled for a early rehabilitation intervention through multisensory stimulations, a rehabilitation specifically aimed at improving the visual field deficit, possibly combined with standard physical rehabilitation in temporary hospitalization facilities or protected hospital discharge.
  Interventions: Other: Early multisensory audio-visual stimulation training; Diagnostic Test: Early visual field test

INTERVENTIONS:
Other: Early multisensory audio-visual stimulation training — Multisensory audio-visual stimulation training (using the device AV DESK Linari Medical) will last four weeks. Through audiovisual stimuli produced by the Av-Desk Flexi device, patients undergo a brain cell training program that compensates for blind spots in their visual field. The recipes regulating the combinations of stimuli are provided daily, under the supervision of a physician, where the data processing unit manages the data from the stimuli provided to the patient, their response to said stimuli, and monitors their position.
  The follow up visual field test will detect whether early intervention with multisensory audio-visual stimuli can improve visual field loss
  Other Names: audio-visual stimulation
  Arms: Early intervention rehabilitation
Diagnostic Test: Early visual field test — Visual field assessment with wearable devices (PalmScan VF2000) performed at the bedside in post-stroke patients who met the inclusion criteria during their stay in the neurology hospital unit, as soon as they were stabilized.
  Standard 120-point visual field tests will be performed on the left and right eyes separately, with the following quantification parameters: test duration, fixation losses, false positives, false negatives, points seen, points not seen, relative defects.
  Patients with a monocular residual perimetric defect of less than 106 points seen out of 124 (equal to 85% of the stimuli presented) and in any case with a defect greater than 12 points if presented in a single quadrant, will be selected for the clinical trial and invited to repeat the same visual field evaluation, using the same wearable devices in the 2-months follow-up.

SUMMARY:
In this study, the investigators will use a wearable device capable of performing this bedside assessment to evaluate the incidence of visual field loss in post-stroke patients. Furthermore, for those with visual field loss, the investigators will investigate whether integrating multisensory audio-visual rehabilitation into the standard physical rehabilitation protocol can help improve visual field loss compared to standard rehabilitation alone.

DETAILED DESCRIPTION:
The objectives of the research are:

1. To quantify the incidence and severity of visual field defects in subjects with a recent cerebrovascular accident admitted to the hospital Neurology Unit
2. To evaluate the rate of spontaneous recovery of visual field defects during observation .
3. To test the effectiveness of an early and intensive visual rehabilitation intervention based on multisensory stimulation in reducing the severity of the aforementioned visual defect.

The research is planned to be conducted in Genova Italy and to include 300 patients.

In this study, the investigators will recruit acute post-stroke patients from the Neurology Unit of IRCCS Policlinico San Martino hospital. The study will use a wearable device (PalmScan VF2000) to assess the visual field defects. Those with significant visual field defects will be randomly assigned to either the visual rehabilitation group, receiving visual rehabilitation treatment integrated into their physical rehabilitation protocol, or the standard group. Inclusion criteria include: age between 18 and 90 years, post-stroke patients (excluding isolated cerebellar, brainstem, or spinal cord strokes), admitted to the Neurology Unit of the IRCCS Policlinico San Martino hospital, able to understand and sign the informed consent for study participation, and having mobility in at least one upper limb. Exclusion criteria include: cognitive impairment that limits understanding of the informed consent or testing, difficulty with both upper limb movements, presence of ocular comorbidity that could affect pre-ictal visual field assessment, presence of fluid aphasia, neglect or deviation of the head and gaze, impaired consciousness or delirium. Baseline assessments will be conducted at the Neurology Unit of the IRCCS Policlinico San Martino hospital.

After the baseline assessment, all participants diagnosed with visual field impairment will be assigned to the David Chiossone Foundation, with the option of being referred to a post-acute residential facility or undergoing outpatient treatment. Otherwise, patients requiring intensive care will be referred to another competent local center.

Participants will be randomly divided into two groups:

* one will receive an early visual rehabilitation protocol (experimental group), possibly supplemented with neuromotor rehabilitation, immediately after discharge from the Neurology Unit of the IRCCS Policlinico San Martino hospital, with a four-week intensive stimulation protocol. Visual rehabilitation will be administered with multisensory audiovisual stimulation (AvDesk) five days a week.
* another group will continue according to current clinical practice (control group), potentially receiving neuromotor rehabilitation until full recovery, and will have access to visual rehabilitation thereafter through the access procedures agreed with the Italian National Health Service.

After 8 weeks since they are dismissed by the hospital Neurology Unit, all patients (even those not receiving vision rehabilitation) will receive a follow-up visual field assessment using the wearable device at the David Chiossone Foundation - for the rehabilitation of blind, visually impaired, and frail people - Social Enterprise.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 99 years with stroke (excluding isolated cerebellar, brainstem, or spinal cord strokes), admitted to Neurology in IRCCS San Martino Polyclinic Hospital with the ability to understand and sign the informed consent for study participation.
2. Mobility of at least one upper limb.

Exclusion Criteria:

1. Presence of cognitive impairment (with an MMSE score less than 24), which limits the understanding of the informed consent or the ability to perform the test.
2. Difficulty moving both upper limbs.
3. Presence of ocular comorbidity that could affect visual field assessment before stroke.
4. Presence of fluent aphasia, neglect, or head and gaze deviation.
5. Presence of disturbances in the state of consciousness
6. Presence of delirium

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Recovery rate in patients who receive training with multisensory audio-visual stimuli | 2 months
  Visual field test (120pt neuro programme) per each eye at follow up compared with the screening test. The functional rate will be in percentage (on 124 stimuli) adding 1 integer for seen points, 0.5 for relative points
Spontaneous recovery rate of visual field defects after stroke | 2 months
  Visual field test (120pt neuro programme) per each eye at follow up compared with the screening test. The functional rate will be in percentage (on 124 stimuli) adding 1 integer for seen points, 0.5 for relative points

SECONDARY OUTCOMES:
Incidence of visual field defects in post-stroke patients | 1 year
  Number of patients with visual field defects, will be compared with literature and retrospective study on clinical records of the hospital neurology clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Schenone, Prof., Principal Investigator — University of Genova DINOGMI

IPD SHARING:
Plan to Share IPD: No